CLINICAL TRIAL: NCT07122518
Title: A Post-Approval Evaluation of the PALMAZ MULLINS XD™ Pulmonary Stent in the Treatment of Pulmonary Artery Stenosis (REALPASS)
Brief Title: Post-Approval Study of PALMAZ MULLINS XD™ in Treating Pulmonary Artery Stenosis
Acronym: REALPASS
Status: Not yet recruiting | Type: Observational
Sponsor: Cordis US Corp. (Industry)
Collaborators: Congenital Cardiovascular Interventional Study Consortium (CCISC) (Unknown)
Responsible Party: Sponsor
Other Study IDs: P23-8501
Record Dates: First submitted 2025-07-02; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Artery Stenosis
Keywords: pulmonary artery stenosis; Pulmonary Artery Stenting; PALMAZ MULLINS XD Pulmonary Stent
MeSH Terms: conditions — Stenosis, Pulmonary Artery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Palmaz Mullins XD™ Treatment: All enrolled subjects are treated with the PALMAZ MULLINS XD™ Pulmonary Stent
  Interventions: Device: PALMAZ MULLINS XD™ Pulmonary Stent

INTERVENTIONS:
Device: PALMAZ MULLINS XD™ Pulmonary Stent — The PALMAZ MULLINS XD™ Pulmonary Stent is indicated for the non-emergency treatment of pulmonary artery stenosis in pediatric patients who are at least 10kg in weight with two ventricle anatomy. The PALMAZ MULLINS XD™ Pulmonary Stent is a balloon-expandable, laser cut stent made from 316L stainless steel tubing. The stent is supplied unmounted and in five (5) nominal unexpanded lengths: 19 mm, 25 mm, 29 mm, 39 mm, and 59 mm.

SUMMARY:
The purpose of the clinical investigation is to characterize clinical outcomes and to assess the real-world use of the commercial PALMAZ MULLINS XD™ Pulmonary Stent.

DETAILED DESCRIPTION:
The clinical study is a prospective, single-arm, multi-center, post-approval study of all consecutive subjects treated with the PALMAZ MULLINS XD™ Pulmonary Stent. The study will enroll a minimum of 35 subjects and a maximum of 75 subjects in up to 11 U.S sites or until the end of the 2-year enrollment period has been reached, whichever comes first.

The study will collect the performance and safety data of the PALMAZ MULLINS XD™ Pulmonary Stent through time of hospital discharge.

ELIGIBILITY:
- Subjects *should* meet criteria as per the list of indications/contraindications in the Instructions for Use, though all subjects treated with PALMAZ MULLINS XD™ Pulmonary Stent will be considered eligible and enrolled.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects with pulmonary artery stenosis who are candidates for treatment with the PALMAZ MULLINS XD™ Pulmonary Stent according to clinical guidelines and/or the operators' judgement will be eligible for enrollment in this study.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Technical Success (Successful use of the study device without additional, unplanned device or procedure-related surgery/re-intervention) | Start time of index procedure through time of discharge/study completion, usually within ~48 hours from end time of index procedure
  1. Successful access, delivery and retrieval of the device delivery system,
  2. Deployment and correct positioning of the device in the intended location, and
  3. No need for additional, unplanned surgery or re-intervention related to the device or access procedure.
Patency (Angiographically-determined increase in stented vessel minimum pulmonary artery diameter by ≥ 50% of the pre-stent diameter) | Index procedure (start time to end time)
  Increase in stented vessel minimum pulmonary artery diameter by ≥ 50% of the pre-stent diameter determined by post-implant angiography.
Safety Outcome (Incidence of Treatment-Emergent Serious Adverse Events) | Time of enrollment (device implant during index procedure) through time of discharge/study completion, usually within ~48 hours from end time of index procedure
  Device or procedure-related, serious adverse events reported through time of hospital discharge, which meet any of the following criteria:
  1. Led to a death,
  2. Led to a serious deterioration in health of the subject, that either resulted in
     1. Life-threatening illness or injury, or
     2. Hospitalization (initial or prolonged) or
     3. Disability or permanent impairment of a body structure or a body function or
     4. Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function
  3. Other Serious (important) Medical Events

OTHER OUTCOMES:
Baseline Characteristics - Demographics | Pre-procedure baseline
  Demographics (age, gender)
Baseline Characteristics - Medical History | Pre-procedure baseline
  Medical History (diagnosis, prior surgery)
Baseline Characteristics - Clinical History: Weight | Pre-procedure baseline
  Clinical History (weight in kg)
Baseline Characteristics - Clinical History: Height | Pre-procedure baseline
  Clinical History (height in cm)
Baseline Characteristics - Clinical History: Body Surface Area | Pre-procedure baseline
  Clinical History (body surface area in square meters)
Target Vessel Characteristics (Stenosis type and location, lesion length and target vessel diameters) | Angiography during index procedure
  Stenosis type and location, lesion length and target vessel diameters
Procedural Characteristics (occurrence and outcomes of pre-dilation, stent deployment and post-dilation during index procedure) | Index procedure
  Occurrence and outcomes of pre-dilation, stent deployment and post-dilation during index procedure
Device Characteristics - Dimensions of PALMAZ MULLINS XD™ Pulmonary Stent | Index procedure
  PALMAZ MULLINS XD™ Pulmonary Stent dimensions
Device Characteristics - Balloon Manufacturer/Model and Dimensions | Index procedure
  Balloon manufacturer/model and dimensions
Device Characteristics - Sheath Manufacturer/Model and Dimensions | Index procedure
  Sheath manufacturer/model and dimensions

IPD SHARING:
Plan to Share IPD: Undecided